CLINICAL TRIAL: NCT01190306
Title: Safety and Effectiveness of the VEGA UV-A System for Corneal Collagen Cross-Linking in Eyes With Keratoconus
Brief Title: Safety Study of the VEGA UV-A System to Treat Keratoconus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor terminated the study prior to data analysis for financial reasons.
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXL-001
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Results first posted 2013-03-04 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CXL Treatment (Experimental): Eyes randomized to the CXL treatment group with be treated with riboflavin and UV light.
  Interventions: Device: The VEGA UV-A Illumination System; Drug: Riboflavin
- Sham Control (Active Comparator): Eyes in the control group will be treated with riboflavin only.
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Device: The VEGA UV-A Illumination System — This is a portable electronic device designed to deliver a dose of UV-A light to the treatment area
  Arms: CXL Treatment
Drug: Riboflavin — Riboflavin is a solution that will be delivered to the treatment area

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of corneal collagen cross-linking (CXL), when used to treat keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older
* Having a diagnosis of keratoconus
* Presence of central or inferior steepening
* Topography consistent with keratoconus
* Presence of one or more slit lamp or retinoscopy findings associated with keratoconus
* Contact lens wearers only:Removal of contact lenses for the required period of time
* Signed written informed consent
* Willingness and ability to comply with schedule for follow-up visits

Exclusion Criteria:

* For keratoconus, a history of previous corneal surgery or the insertion of Intacs in the eye to be treated
* Corneal pachymetry ≤ 400 microns
* Previous ocular condition that may predispose the eye for future complications or prevent the possibility of improved vision
* A history of chemical injury or delayed epithelial healing in the eye(s) to be treated.
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Nystagmus or any other condition that would prevent a steady gaze during the cross-linking treatment or other diagnostic tests
* A condition that, in the investigator's opinion, would interfere with or prolong epithelial healing.
* Presence or history of any other condition or finding that, in the investigator's opinion, makes the patient unsuitable as a candidate for cross-linking or study participation or may confound the outcome of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Woolfson Eye Institute, Atlanta, Georgia
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - Pamel Vision & Laser Group, New York, New York
  - Mt. Sinai Hospital, New York, New York
  - OSU Department of Ophthalmoloty, Columbus, Ohio
  - Revision Advanced Laser Eye Center, Columbus, Ohio
  - Dell Laser Consultants, Austin, Texas
  - Slade & Baker Vision Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from August, 2010 to December 2011 from medical clinics throughout the country.
Pre-assignment Details: Patients that were excluded from the clinical trial were considered screen failures due to not meeting one or more of the inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | CXL Treatment | Sham Control
Started | 61 | 66
Completed | 61 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CXL Treatment | Sham Control | Total
Number analyzed (Participants) | 61 | 66 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — The sponsor terminated the study prior to data analysis for financial reasons. | NA — The sponsor terminated the study prior to data analysis for financial reasons. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | NA — The sponsor terminated the study prior to data analysis for financial reasons. | NA — The sponsor terminated the study prior to data analysis for financial reasons. | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — The sponsor terminated the study prior to data analysis for financial reasons. | NA — The sponsor terminated the study prior to data analysis for financial reasons. | NA — Total not calculated because data are not available (NA) in one or more arms.
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — The sponsor terminated the study prior to data analysis for financial reasons. | NA (NA) — The sponsor terminated the study prior to data analysis for financial reasons. | NA (NA) — The sponsor terminated the study prior to data analysis for financial reasons.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — The sponsor terminated the study prior to data analysis for financial reasons. | NA — The sponsor terminated the study prior to data analysis for financial reasons. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — The sponsor terminated the study prior to data analysis for financial reasons. | NA — The sponsor terminated the study prior to data analysis for financial reasons. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | NA — The sponsor terminated the study prior to data analysis for financial reasons | NA — The sponsor terminated the study prior to data analysis for financial reasons | NA — The sponsor terminated the study prior to data analysis for financial reasons

OUTCOME MEASURES:

1. Primary Outcome: Change in Corneal Curvature.
Time Frame: 6 Months
Population: The CXL-001 study was completed but data analysis was not done. Prior to data analysis, the sponsor, Topcon, decided to terminate the study for administrative reasons only, and not as a result of any safety issues or concerns relating to the study.
Arm/Group | CXL Treatment | Sham Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | CXL Treatment | Sham Control
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/66
Other Adverse Events (participants affected / at risk) | 0/61 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All such Confidential Information shall remain the property of Topcon, as applicable, and Institution agrees that neither it nor Principal Investigator nor any of its employees or Sub-Investigators, if any, shall disclose any of the Confidential Information to third parties, without the prior written consent of Topcon.